CLINICAL TRIAL: NCT07210619
Title: Expanded Access for d-MAPPS™ Ophthalmic Solution, in the Treatment of Chronic Ocular Graft-Versus-Host Disease (oGVHD)
Status: Available | Type: Expanded Access
Sponsor: Regenerative Ocular Immunobiologics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 30066-EA
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: oGVHD

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: d-MAPPS — Ophthalmic Solution for oGVHD

SUMMARY:
Regenerative Ocular Immunobiologics, LLC Fast Track Expanded Access This Expanded Access Policy describes the conditions under which ROI may make its investigational product - Sterile Processed Derived Multiple Allogeneic Proteins Paracrine Signaling (d-MAPPS™ Ophthalmic Solution) - available to patients outside of a clinical trial, in accordance with U.S. FDA regulations, including section 561A of the Federal Food, Drug, and Cosmetic Act (FDCA).

DETAILED DESCRIPTION:
Regenerative Ocular Immunobiologics, LLC ("ROI") is committed to advancing innovative regenerative biologics for serious ocular conditions with high unmet medical need. The investigational product, d-MAPPS™ Ophthalmic Solution, is currently being evaluated in clinical trials under U.S. FDA Investigational New Drug (IND) #030066. Clinical trial participation remains the preferred and primary pathway for patient access. ROI has established this Expanded Access Policy in accordance with Section 561A of the FDCA to outline conditions under which d-MAPPS™ may be considered outside of a clinical trial.

At this stage of development, d-MAPPS™ is not approved by the FDA. Participation in a clinical trial is the preferred mechanism for accessing this investigational treatment, as trials are designed to evaluate safety and effectiveness in a controlled setting.

Certain patients with serious or immediately life-threatening conditions may not meet eligibility criteria for clinical trials and may pursue access to investigational therapies. In accordance with Section 561A of the Federal Food, Drug, and Cosmetic Act, Regenerative Ocular Immunobiologics has established the following Expanded Access (EA) policy:

This Expanded Access Policy describes the conditions under which Sterile Processed Derived Multiple Allogeneic Proteins Paracrine Signaling (d-MAPPS™ Ophthalmic Solution) may be made available to patients outside of a clinical trial, in accordance with U.S. FDA regulations.

Availability

* Expanded Access to d-MAPPS™ may be considered for patients with severe chronic ocular GVHD who have no satisfactory alternative treatment options and who are not eligible for ongoing clinical trials.
* Expanded Access is not guaranteed and remains subject to review of patient circumstances, clinical data, and drug supply.

Request Procedures Treating ophthalmologists or eye care professionals may submit Expanded Access requests to info@roiglobalsolutions.org.

Requests should include relevant patient history, diagnosis, rationale for Expanded Access, and a proposed monitoring plan.

Criteria for Consideration

Requests will be evaluated on the following:

* Seriousness of the patient's condition
* Lack of satisfactory therapeutic alternatives
* Ineligibility for ongoing clinical trials
* Whether potential benefit justifies potential risk of the investigational product
* Adequate drug supply

Review and Response Timeline Regenerative Ocular Immunobiologics will acknowledge receipt of EA requests within 5 business days and will provide a decision as promptly as possible while following all FDA requirements. All requests will be reviewed in accordance with FDA regulations and company policy.

Cost of Treatment ROI does not currently intend to charge patients for d-MAPPS™ provided through Expanded Access. ROI reserves the right to recover direct costs in accordance with FDA regulations should circumstances change.

Policy Updates

This Expanded Access Policy will be reviewed and updated as needed. The most current version will be available at:

https://www.roiglobalsolutions.org/

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Willing and able to provide written informed consent.
* Willing and able to comply with study assessments for the full duration of the study.
* Patients may be using bilateral scleral lenses and/or bilateral punctal plugs at the time of accrual.
* Minimum Oxford Schema grade of ≥1 in at least one eye.
* OSDI score of ≥22.
* UNC DEMS score of ≥3.
* In good stable overall health
* Note: If the patient has no exclusion criteria, investigator can combine the Pre-screen and Baseline visit

Exclusion Criteria:

* History of Rheumatoid Arthritis, Lupus, Scleroderma. (Exception may be made at the discretion of the Principal Investigator if it is determined that the patient would benefit from d-MAPPS ophthalmic solution).
* Ocular or periocular malignancy.
* Significant change, as judged by the principal investigator, in systemic immunosuppressive regimen within 2 weeks of study entry.
* Any history of topical tacrolimus use (Exception may be made at the discretion of the Principal Investigator if it is determined that the patient would benefit from d-MAPPS ophthalmic solution).
* Any change in dosage of tetracycline compounds (tetracycline, doxycycline, and minocycline) within the last month.
* Any change in frequency of preserved anti-glaucoma medications within 2 weeks of study entry.
* Current use of topical steroids more than twice a day.
* Corneal epithelial defect >1mm2.
* Any history of herpetic keratitis. (Exception may be made at the discretion of the Principal Investigator if it is determined that the patient would benefit from d-MAPPS ophthalmic solution).
* Participation in another simultaneous medical research study.
* Signs of current infection, including fever and current treatment with antibiotics.
* All vaccinations including COVID are prohibited during this study.
* Intra-ocular surgery or ocular laser surgery within 3 months. (Exception may be made at the discretion of the Principal Investigator if it is determined that the patient would benefit from d-MAPPS ophthalmic solution following surgery.)
* Women who are pregnant, breastfeeding, or plan to become pregnant while participating in the study. If of child-bearing potential, unwillingness to use effective birth control while participating in the study.)
* Any condition (including language barrier) that precludes patient's ability to comply with study requirements including completion of study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- See also: Website for ROI Global — https://www.roiglobalsolutions.org/